CLINICAL TRIAL: NCT04443634
Title: Presurgical Adductor Canal Block (ACB) Versus ACB and Distal (Intermuscular) Saphenous Nerve Block in Patients Undergoing Anterior Cruciate Ligament Repair Under General Anaesthesia: Randomised Controlled Trial.
Brief Title: Adductor Canal Block (ACB) Versus ACB /Saphenous Block in Patients Undergoing Anterior Cruciate Ligament Repair
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Bassant M. Abdelhamid, associate professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: N-27-2017
Record Dates: First submitted 2020-06-18; First posted 2020-06-23 (Actual); Last update posted 2020-06-29 (Actual); Status verified 2020-06

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Anesthesia, General; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Adductor 20 (Experimental): Ultrasound guided adductor canal block will be performed with injection of 20 ml bupivacaine
  Interventions: Procedure: Ultrasound Guided Adductor Canal Block; Procedure: General anesthesia; Drug: Bupivacaine 20 ml
- Adductor 30 (Experimental): Ultrasound guided adductor canal block will be performed with injection of 30ml bupivacaine
  Interventions: Procedure: Ultrasound Guided Adductor Canal Block; Procedure: General anesthesia; Drug: Bupivacaine 30ml
- Adductor /Saphenous (Experimental): Ultrasound guided adductor canal block will be performed by injection of 20 ml bupivacaine , combined with ultrasound guided saphenous nerve block at the distal third of the thigh in the intermuscular plane between Vastus Medialis and Sartorius muscle with injection of 10ml bupivacaine 0.5%.
  Interventions: Procedure: Ultrasound Guided Adductor Canal Block; Procedure: Ultrasound Guided Saphenous Nerve Block; Procedure: General anesthesia; Drug: Bupivacaine 20 ml; Drug: Bupivacaine 10ml

INTERVENTIONS:
Procedure: Ultrasound Guided Adductor Canal Block — It will be performed at the midthigh level, approximately halfway between the superior anterior iliac spine and the patella, a high-frequency linear ultrasound (US) transducer 5-12 MHz probe. Underneath the sartorius muscle the femoral artery was identified, with the vein just inferior and the saphenous nerve just lateral to the artery. From the lateral side of the transducer a 10-cm, 18-gauge Tuohy needle (Braun Medical, Melsungen, Germany) was inserted in plane, through the Sartorius muscle. With the tip of the Tuohy needle placed just underneath the vasto-adductor membrane and lateral to the artery and the saphenous nerve, 20 ml local anesthetic mixture will be injected to expand the adductor canal. the volume of local anesthetic will be selected according to the studied group
Procedure: Ultrasound Guided Saphenous Nerve Block — It will be performed at the intermuscular plane between the sartorius and the vasus medialis muscles at the lower third of the thigh.
  The US probe will be positioned on the front of the lower part of the thigh immediately above the patella to see both the patella (hyperechoic curved line) and vastus medialis infront of it (closer to skin). The probe is then moved medially over the vastus medialis till we see the end of the muscle and we see an intermuscular plane between it and Sartorius muscle. A 20 guage spinal needle will be then passed in an in plane direction within the substance of vastus medialis muscle and then pass within the vastus medialis until it faces the intermuscular plane between VM muscle and Sartorius. Once the needle tip is located in close proximity to the target structures, gentle aspiration will be performed followed by 20 ml local anesthetic will be injected.
  Arms: Adductor /Saphenous
Procedure: General anesthesia — General anesthesia was induced by propofol 1-2 mg/kg fentanyle 100micg and laryngeal mask was inserted. Maintanace of anesthesia was performed by sevoflurane 2-3%.
  Then the surgical procedure started. All patients had arthroscopic knee surgery( ACL repair) surgery under tourniquet control.
  Immediately after end the surgical procedure, either ACB or combined ACB and saphenous nerve block distal to adductor canal were performed according to randomization.
Drug: Bupivacaine 20 ml — 20ml bupivacaine 0.5%
  Arms: Adductor /Saphenous; Adductor 20
Drug: Bupivacaine 30ml — 30ml bupivacaine 0.5%
  Arms: Adductor 30
Drug: Bupivacaine 10ml — 10ml bupivacaine 0.5%
  Arms: Adductor /Saphenous

SUMMARY:
Knee surgeries are associated with severe postoperative pain. Blocking the femoral nerve (or saphenous nerve) in the adductor canal is increasingly used for knee analgesia. It carries potential benefits that encourage anesthesiologists to do it. It has a motor sparing property. Injection of local anesthetics in this lengthy canal that contains a variable amount of connective or fibrous tissue might lead to a patchy distribution of local anesthetics. Thus, the possibility of incomplete block of the saphenous nerve (most important nerve in knee innervations) cannot be excluded.

DETAILED DESCRIPTION:
Aim of the study is to compare the efficacy of the adductor canal block to the combined adductor canal block and saphenous nerve block at the distal third of thigh in the intermuscular plane between Vastus Medialis and Sartorius muscles in pain relief following knee arthroscopic anterior cruciate ligament repair.

After written informed consent, patients will be randomized in three groups:

Group (Adductor 20): Ultrasound guided adductor canal block will be performed with injection of 20 ml bupivcaine 0.5%.

Group (Adductor 30) Ultrasound guided adductor canal block will be performed with injection of 30 ml bupivacaine 0.5%. Group (Adductor/saphenous ): Ultrasound guided adductor canal block will be performed by injection of 20 ml bupivacaine 0.5%, combined with ultrasound guided saphenous

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for knee orthopedic ( ACL repair)
* Physical status ASA I, II.
* Body mass index (BMI): > 20 kg/m2 and < 35 kg/m2.

Exclusion Criteria:

* • Patients with known sensitivity or contraindication to drug used in the study (local anesthetics, opioids).

  * History of psychological disorders and/or chronic pain.
  * Contraindication to regional anesthesia e.g. local sepsis, pre- existing peripheral neuropathies and coagulopathy.
  * Infection of the skin at the site of needle puncture area.
  * Patient refusal.
  * Severe respiratory or cardiac disorders.
  * Advanced liver or kidney disease.
  * Pregnancy.
  * Patient with surgery duration more than two hours.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2020-06-25 (Actual); Primary Completion 2020-09-25 (Estimated); Study Completion 2020-10-01 (Estimated)

PRIMARY OUTCOMES:
The total dose of morphine consumption in the first 24 hours postoperatively. | 24 hours postoperative
  The total amount of morphine consumption in the first 24 hours postoperatively.

SECONDARY OUTCOMES:
Total dose of intraoperative fentanyle adminstration | 2 hours intraoperatively
Numeric Pain Rating Scale | 24 hours postoperative
  Numeric Pain Rating Scale, both at rest and during movement: 30 minutes,2, 4,6, 8, 12, 16, 20 and 24 hours postoperatively. It is labeled from zero to ten, with zero being an example of someone with no pain and ten being the worst pain possible.
Failure rate of the block | 24 hours
  • Failure rate of the block will be calculated, where the block will be considered a failed block if the patient requires more than two doses of rescue analgesia in the first hour postoperatively.
Block related complications | 1 mounth
  o The incidence of vascular puncture, and presence or absence of saphenous nerve neuritis during the first month after surgery were also recorded

CONTACTS AND LOCATIONS:
Overall Officials: Bassant abdelhamid, Principal Investigator — Cairo University
Locations (1):
- Anesthesia Department, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ilfeld BM, Duke KB, Donohue MC. The association between lower extremity continuous peripheral nerve blocks and patient falls after knee and hip arthroplasty. Anesth Analg. 2010 Dec;111(6):1552-4. doi: 10.1213/ANE.0b013e3181fb9507. Epub 2010 Oct 1. PMID 20889937
- [Background] Ilfeld BM, Moeller LK, Mariano ER, Loland VJ, Stevens-Lapsley JE, Fleisher AS, Girard PJ, Donohue MC, Ferguson EJ, Ball ST. Continuous peripheral nerve blocks: is local anesthetic dose the only factor, or do concentration and volume influence infusion effects as well? Anesthesiology. 2010 Feb;112(2):347-54. doi: 10.1097/ALN.0b013e3181ca4e5d. PMID 20098137
- [Background] Jaeger P, Koscielniak-Nielsen ZJ, Schroder HM, Mathiesen O, Henningsen MH, Lund J, Jenstrup MT, Dahl JB. Adductor canal block for postoperative pain treatment after revision knee arthroplasty: a blinded, randomized, placebo-controlled study. PLoS One. 2014 Nov 11;9(11):e111951. doi: 10.1371/journal.pone.0111951. eCollection 2014. PMID 25386752
- [Background] Manickam B, Perlas A, Duggan E, Brull R, Chan VW, Ramlogan R. Feasibility and efficacy of ultrasound-guided block of the saphenous nerve in the adductor canal. Reg Anesth Pain Med. 2009 Nov-Dec;34(6):578-80. doi: 10.1097/aap.0b013e3181bfbf84. PMID 19916251